CLINICAL TRIAL: NCT02164253
Title: Feasibility and Safety Pilot Therapeutic Study of the Iron Chelator Deferiprone in Amyotrophic Lateral Sclerosis
Brief Title: Focal Accumulation of Iron in Cerebral Regions in Early ALS (Amyotrophic Lateral Sclerosis) Patients
Acronym: SAFEFAIRALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012_69; 2013-001228-21 (EudraCT Number)
Record Dates: First submitted 2014-05-20; First posted 2014-06-16 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2016-10

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis); Iron Overload
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Iron Overload | interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferiprone (Experimental): Deferiprone, 25 to 30 mg/kg per day, oral use
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone — 30 mg/kg per day, oral use
  Other Names: Ferriprox

SUMMARY:
The FAIR-ALS study is to investigate the safety and efficacy of a scavenger treatment of iron deferiprone, which would reduce the brain iron to limit the development of amyotrophic lateral sclerosis.

It has been shown an excess of iron in the central nervous system carrying a sporadic ALS patients. Iron overload associated with a loss of motor neurons may explain the signs of the disease (atrophy).

The investigators discuss the hypothesis that reducing excess iron, the investigators can reduce the loss of neurons and thus the progression of signs of the disease.

DETAILED DESCRIPTION:
At the end of the study, it will propose to continue the usual quarterly patient follow up, as recommended by the French ALS centers.

Deferiprone can be administered as part of a compassionate use, for patients who want it and who do not have hypoxemia.

We therefore plan a treatment period compassionate relatively short and less than 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic lateral sclerosis defined in accordance to the El Escorial criteria (possible, probable or defined)
* 18 to 85 years old patient, male or female
* Patient with social security cover

Exclusion Criteria:

* Achieved respiratory defined by a FVC <70%
* Evolution of more than 24 months
* Demented subject
* Severe malnutrition
* Patients with treatment potentially at risk of agranulocytosis and neutropenia
* Patients with a history of agranulocytosis or iatrogenic under haematological disease
* Incapable of giving consent
* Indication against MRI
* Indication against lumbar puncture
* Patient refused lumbar puncture
* Hypersensitivity to iron chelators
* Concomitant treatment with antacids containing aluminum
* Presence of another serious illness to life-threatening or disabling cons to the use of the treatment mixture of oxygen and nitrous oxide equally

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evolution of Amyotrophic Lateral Sclerosis Functional Rating Scale | V3, V6, V9, V12, V15

SECONDARY OUTCOMES:
Comparison of the progression of ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale ) score for 3 months without treatment (V0 to V3) in the period of the first three months under treatment (V3 to V6). | SCREENING, V0, V3, V6
The proportion of patients who become non-self-sufficient after 12 months with the appearance of a sub scores ALSFRS-R less than or equal to 2 on swallowing, cut food using utensils or walk. | SCREENING, V0, V3, V6, V9, V12, V15
Number of patients with anemia at 12 months defined by a hemoglobin / dL Hb <12 g | V3, V6, V9, V12, V15
Number of serious and non-serious adverse events | SCREENING, V0, V3, V6, V9, V12, V15
Progression of respiratory vital capacity tests | SCREENING, V0, V3, V6, V9, V12, V15
Values of R2 * in MRI | V3, V6, V19
Oxidative stress markers analyzed blindly in blood and cerebrospinal fluid | V3, V9
No alteration of energy metabolism in aerobic and anaerobic blood and cerebrospinal fluid | V3, V9

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Moreau, MD, Principal Investigator — UH Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

REFERENCES:
- [Background] Bensimon G, Lacomblez L, Meininger V. A controlled trial of riluzole in amyotrophic lateral sclerosis. ALS/Riluzole Study Group. N Engl J Med. 1994 Mar 3;330(9):585-91. doi: 10.1056/NEJM199403033300901. PMID 8302340
- [Background] Boddaert N, Le Quan Sang KH, Rotig A, Leroy-Willig A, Gallet S, Brunelle F, Sidi D, Thalabard JC, Munnich A, Cabantchik ZI. Selective iron chelation in Friedreich ataxia: biologic and clinical implications. Blood. 2007 Jul 1;110(1):401-8. doi: 10.1182/blood-2006-12-065433. Epub 2007 Mar 22. PMID 17379741
- [Background] Danzeisen R, Achsel T, Bederke U, Cozzolino M, Crosio C, Ferri A, Frenzel M, Gralla EB, Huber L, Ludolph A, Nencini M, Rotilio G, Valentine JS, Carri MT. Superoxide dismutase 1 modulates expression of transferrin receptor. J Biol Inorg Chem. 2006 Jun;11(4):489-98. doi: 10.1007/s00775-006-0099-4. Epub 2006 Apr 26. PMID 16680451
- [Background] Felice KJ. A longitudinal study comparing thenar motor unit number estimates to other quantitative tests in patients with amyotrophic lateral sclerosis. Muscle Nerve. 1997 Feb;20(2):179-85. doi: 10.1002/(sici)1097-4598(199702)20:23.0.co;2-9. PMID 9040656
- [Background] Goodall EF, Greenway MJ, van Marion I, Carroll CB, Hardiman O, Morrison KE. Association of the H63D polymorphism in the hemochromatosis gene with sporadic ALS. Neurology. 2005 Sep 27;65(6):934-7. doi: 10.1212/01.wnl.0000176032.94434.d4. PMID 16186539
- [Background] Kwiatkowski A, Ryckewaert G, Jissendi Tchofo P, Moreau C, Vuillaume I, Chinnery PF, Destee A, Defebvre L, Devos D. Long-term improvement under deferiprone in a case of neurodegeneration with brain iron accumulation. Parkinsonism Relat Disord. 2012 Jan;18(1):110-2. doi: 10.1016/j.parkreldis.2011.06.024. Epub 2011 Aug 6. No abstract available. PMID 21821461
- [Background] Kong J, Xu Z. Massive mitochondrial degeneration in motor neurons triggers the onset of amyotrophic lateral sclerosis in mice expressing a mutant SOD1. J Neurosci. 1998 May 1;18(9):3241-50. doi: 10.1523/JNEUROSCI.18-09-03241.1998. PMID 9547233
- [Background] Langkammer C, Enzinger C, Quasthoff S, Grafenauer P, Soellinger M, Fazekas F, Ropele S. Mapping of iron deposition in conjunction with assessment of nerve fiber tract integrity in amyotrophic lateral sclerosis. J Magn Reson Imaging. 2010 Jun;31(6):1339-45. doi: 10.1002/jmri.22185. PMID 20512885
- [Background] Lin J, Diamanduros A, Chowdhury SA, Scelsa S, Latov N, Sadiq SA. Specific electron transport chain abnormalities in amyotrophic lateral sclerosis. J Neurol. 2009 May;256(5):774-82. doi: 10.1007/s00415-009-5015-8. Epub 2009 Feb 25. PMID 19240958
- [Background] Miller R, Bradley W, Cudkowicz M, Hubble J, Meininger V, Mitsumoto H, Moore D, Pohlmann H, Sauer D, Silani V, Strong M, Swash M, Vernotica E; TCH346 Study Group. Phase II/III randomized trial of TCH346 in patients with ALS. Neurology. 2007 Aug 21;69(8):776-84. doi: 10.1212/01.wnl.0000269676.07319.09. PMID 17709710
- [Background] Moreau C, Gosset P, Kluza J, Brunaud-Danel V, Lassalle P, Marchetti P, Defebvre L, Destee A, Devos D. Deregulation of the hypoxia inducible factor-1alpha pathway in monocytes from sporadic amyotrophic lateral sclerosis patients. Neuroscience. 2011 Jan 13;172:110-7. doi: 10.1016/j.neuroscience.2010.10.040. Epub 2010 Oct 25. PMID 20977930
- [Background] Moreau C, Devos D, Gosset P, Brunaud-Danel V, Tonnel AB, Lassalle P, Defebvre L, Destee A. [Mechanisms of deregulated response to hypoxia in sporadic amyotrophic lateral sclerosis: a clinical study]. Rev Neurol (Paris). 2010 Mar;166(3):279-83. doi: 10.1016/j.neurol.2009.05.018. Epub 2009 Aug 5. French. PMID 19660777
- [Background] Moreau C, Gosset P, Brunaud-Danel V, Lassalle P, Degonne B, Destee A, Defebvre L, Devos D. CSF profiles of angiogenic and inflammatory factors depend on the respiratory status of ALS patients. Amyotroph Lateral Scler. 2009 Jun;10(3):175-81. doi: 10.1080/17482960802651725. PMID 19177252
- [Background] Moreau C, Devos D, Brunaud-Danel V, Defebvre L, Perez T, Destee A, Tonnel AB, Lassalle P, Just N. Paradoxical response of VEGF expression to hypoxia in CSF of patients with ALS. J Neurol Neurosurg Psychiatry. 2006 Feb;77(2):255-7. doi: 10.1136/jnnp.2005.070904. PMID 16421133
- [Background] Moreau C, Devos D, Brunaud-Danel V, Defebvre L, Perez T, Destee A, Tonnel AB, Lassalle P, Just N. Elevated IL-6 and TNF-alpha levels in patients with ALS: inflammation or hypoxia? Neurology. 2005 Dec 27;65(12):1958-60. doi: 10.1212/01.wnl.0000188907.97339.76. PMID 16380619
- [Background] Noto Y, Misawa S, Kanai K, Shibuya K, Isose S, Nasu S, Sekiguchi Y, Fujimaki Y, Nakagawa M, Kuwabara S. Awaji ALS criteria increase the diagnostic sensitivity in patients with bulbar onset. Clin Neurophysiol. 2012 Feb;123(2):382-5. doi: 10.1016/j.clinph.2011.05.030. Epub 2011 Jul 20. PMID 21764635
- [Background] Schrooten M, Smetcoren C, Robberecht W, Van Damme P. Benefit of the Awaji diagnostic algorithm for amyotrophic lateral sclerosis: a prospective study. Ann Neurol. 2011 Jul;70(1):79-83. doi: 10.1002/ana.22380. Epub 2011 Mar 17. PMID 21437935
- [Background] Shefner JM, Cudkowicz ME, Zhang H, Schoenfeld D, Jillapalli D; Northeast ALS Consortium. Revised statistical motor unit number estimation in the Celecoxib/ALS trial. Muscle Nerve. 2007 Feb;35(2):228-34. doi: 10.1002/mus.20671. PMID 17058270
- [Background] Shefner JM, Watson ML, Simionescu L, Caress JB, Burns TM, Maragakis NJ, Benatar M, David WS, Sharma KR, Rutkove SB. Multipoint incremental motor unit number estimation as an outcome measure in ALS. Neurology. 2011 Jul 19;77(3):235-41. doi: 10.1212/WNL.0b013e318225aabf. Epub 2011 Jun 15. PMID 21676915
- [Background] Yuen EC, Olney RK. Longitudinal study of fiber density and motor unit number estimate in patients with amyotrophic lateral sclerosis. Neurology. 1997 Aug;49(2):573-8. doi: 10.1212/wnl.49.2.573. PMID 9270599
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820